CLINICAL TRIAL: NCT04348500
Title: A Phase II Trial to Evaluate the Safety and Tolerability of Clazakizumab® (Anti-IL-6 Monoclonal) Compared to Placebo for the Treatment of COVID-19 Infection
Brief Title: Clazakizumab (Anti-Interleukin 6 (IL-6) Monoclonal) Compared to Placebo for Coronavirus Disease 2019 (COVID-19)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Stanley Jordan, MD, Director of Nephrology and Transplant Immunology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00000644
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Results first posted 2021-12-02 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — clazakizumab

STUDY DESIGN:
Intervention Model Description: We propose the administration of a blinded dose of an investigational product (IP) (clazakizumab or placebo [0.9% saline]) in patients with COVID-19 disease and signs of pulmonary involvement who have not yet required mechanical ventilation and/or ECMO. If a patient progresses to mechanical ventilation and/or ECMO or develops clinical signs of deteriorating COVID-19 disease, and there are no treatment related serious adverse events (SAEs), within the initial 14 day period after the first dose of the IP, at the discretion of the investigator or treating physician, open-label clazakizumab 25mg IV x 1 dose may be administered. A minimum of 24 hours should elapse between the first dose of IP and this dose of open-label clazakizumab. The patient will remain blinded as to the identity of the IP administered in the first dose.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded IP (clazakizumab or placebo) will be given initially, followed by the option of an open label dose of clazakizumab within the first 14 days of initial IP administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clazakizumab (Active Comparator): 25 mg in 50 mL of 0.9% saline given by IV infusion x 1 dose over 30 minutes
  Interventions: Drug: Clazakizumab
- Placebo (Placebo Comparator): 50 mL of 0.9% saline given by IV infusion x 1 dose over 30 minutes
  Interventions: Drug: Clazakizumab

INTERVENTIONS:
Drug: Clazakizumab — IV Infusion

SUMMARY:
This is a single center, randomized, double-blind, placebo-controlled, exploratory phase II study enrolling 60 patients. We propose the administration of a blinded dose of an investigational product (IP) (clazakizumab or placebo [0.9% saline]) in patients with COVID-19 disease and signs of pulmonary involvement who have not yet required mechanical ventilation and/or extracorporeal membrane oxygenation (ECMO). If a patient progresses to mechanical ventilation and/or ECMO or develops clinical signs of deteriorating COVID-19 disease, and there are no treatment related serious adverse events (SAEs), within the initial 14 day period after the first dose of the IP, at the discretion of the investigator or treating physician, open-label clazakizumab 25mg IV x 1 dose may be administered. A minimum of 24 hours should elapse between the first dose of IP and this dose of open-label clazakizumab. The patient will remain blinded as to the identity of the IP administered in the first dose.

DETAILED DESCRIPTION:
Patients admitted to the hospital with COVID-19 disease with signs of pulmonary involvement will be randomized to receive the anti-IL-6 drug clazakizumab 25mg IV or placebo. Patients will be followed for improvements in clinical symptoms and laboratory parameters which are part of our COVID-19 lab panel described below. Patients will receive standard of care (SOC) supportive treatment and will be followed for 14 days. If a patient from either group progresses to the need for mechanical ventilation and/or ECMO, or develops clinical signs of deteriorating COVID-19 disease, and there are no serious treatment related SAEs, at the discretion of the investigator or treating physician, the patient may receive a single dose of open-label clazakizumab 25mg IV. A minimum of 24 hours should elapse between the first dose of IP and this dose of open-label clazakizumab.

Enrolled patients will receive clazakizumab 25 mg or placebo (0.9% saline) given by IV infusion over 30 minutes. Clazakizumab will be administered in 50 mL of 0.9% saline on Day 1. COVID-19 lab panel and clinical parameters will be monitored to determine if patients are progressing towards need for ventilation and/or ECMO. The parameters below will be monitored and patient status will be assessed by the clinical team.

If patients do develop these criteria, open-label clazakizumab 25 mg IV may be administered as discussed above. A minimum of 24 hours should elapse between the first dose of IP and this dose of open-label clazakizumab. Patients ventilated with or without ECMO will continue to be monitored post-treatment for signs of improvement, (i.e., decreasing FiO2 requirements, chest X-ray (CXR) improvements, C-reactive protein (CRP) reductions, extubation and discharge home) or death.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 at the time of screening
* Subject must be able to understand and provide informed consent
* Hospitalized with COVID-19 (+) disease (confirmed by polymerase chain reaction (PCR) assay from any specimen (e.g. respiratory, blood, urine, stool, other bodily fluid))
* Not on mechanical ventilation and/or ECMO
* Evidence of pulmonary involvement with at least 2 of the following:

  1. Oxygen saturation (SpO2) at rest in ambient air with SpO2 ≤ 94%
  2. Tachypnea with resting respiration rate > 25 breaths/minute
  3. Partial pressure of oxygen (PaO2) / fraction of inspired oxygen (FiO2) ≤ 300 mmHg
  4. Chest imaging (radiograph, CT scan, or lung ultrasound) with abnormalities consistent COVID-19 pneumonia
  5. C-reactive protein (CRP) >35 mg/L

Exclusion Criteria:

* Previous hypersensitivity or allergic reactions to clazakizumab
* Lactating or pregnant females
* Subjects with latent Tuberculosis (TB) and who are not receiving treatment
* Subjects with active TB
* A significantly abnormal general serum screening lab result defined as a White Blood Count (WBC) < 3.0 X 103/ml, a Hgb < 8.0 g/dL, a platelet count < 50 X 103/ml, a serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) > 5x upper limit normal
* Participation in another clinical trial investigating COVID-19 aimed agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients eligible for the study and who may benefit from the administration of clazakizumab will be identified by members of the inpatient team and referred to the study team. If a patient is eligible, the PI or Co-I will discuss the study with them. Treating physicians of COVID-19 patients will be made aware of the research offering. Patients will be asked if they can be approached about research options. Researchers may approach potential subjects who indicate they are interested.
Pre-assignment Details: Of the total 105 participants ages 18 years and older screened, 17 were enrolled in this single center, randomized, double-blind, placebo-controlled, exploratory phase II study.
Period: Overall Study
Arm/Group | Clazakizumab | Placebo
Started | 8 | 9
Treated | 8 | 8
Completed | 6 | 6
Not Completed | 2 | 3
Not completed — Death | 2 | 2
Not completed — Withdrawn by subject due to dementia | 0 | 1

BASELINE CHARACTERISTICS:
Population: Enrolled patients who received the initial dose of the IP were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Clazakizumab | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (13.44) | 60 (13.14) | 59 (13.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety of Clazakizumab for the Treatment of Patients With COVID-19 Disease
Description: Number of severe adverse events (SAEs) that are unusual, unexpected, or assessed as related to the investigational product (IP)
Time Frame: 14 days
Population: Enrolled patients who received the initial dose of the IP were analyzed.
Measure: Number; unit: Adverse Events
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 8 | 8
Adverse Events
  SAEs within 14 days | 3 | 3
  Adverse Events (AEs) and SAEs overall | 6 | 8
Statistical Analysis 1: Comparison: Clazakizumab vs Placebo; The null hypothesis is that there is no difference in the use of clazakizumab as a treatment compared to placebo in reducing or eliminating the incidence of severe adverse events among patients with COVID-19; Test type: Superiority; p = 0.10, Chi-squared — P-value was not adjusted

2. Secondary Outcome: Patient Survival at 28 Days
Description: Number of patients alive at 28 days
Time Frame: 28 days
Population: Enrolled patients who received the initial dose of the IP were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 7 | 7

3. Secondary Outcome: Patient Survival at 60 Days
Description: Number of patients alive at 60 days
Time Frame: 60 days
Population: Enrolled patients who received the initial dose of the IP were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 6 | 6

4. Secondary Outcome: Number of Patients Requiring the Dose of Open-label Clazakizumab
Description: Number of patients requiring the dose of open-label clazakizumab
Time Frame: 14 days
Population: Enrolled patients who received the initial dose of the IP were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 2 | 5

5. Secondary Outcome: Number of Days in Intensive Care Unit (ICU)
Description: Number of days in ICU compared to placebo
Time Frame: 60 days
Population: Enrolled patients who received the initial dose of the IP were analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 8 | 8
Days | 30.5 (34.65) | 11.67 (3.06)

6. Secondary Outcome: Number of Days in Hospital
Description: Number of days in hospital compared to placebo
Time Frame: 60 days
Population: Enrolled patients who received the initial dose of the IP were analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 8 | 8
Days | 17.5 (16.62) | 18.75 (13.60)

7. Secondary Outcome: Number of Patients Requiring Mechanical Ventilation and/or Extracorporeal Membrane Oxygenation (ECMO)
Description: Number of patients requiring mechanical ventilation and/or ECMO at 14 days after the first administered dose in comparison to placebo
Time Frame: 14 days
Population: Enrolled patients who received the initial dose of the IP were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clazakizumab | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 1 | 2
Statistical Analysis 1: Comparison: Clazakizumab vs Placebo; Null hypothesis is that there is no change in the need for mechanical ventilation and/or ECMO at 14 days after the first administered dose in comparison to placebo; Test type: Superiority; p = 0.10, Fisher Exact — P-value was not adjusted

ADVERSE EVENTS:
Time Frame: Day 60
Description: Enrolled patients who received the initial dose of the IP were monitored and evaluated for adverse and severe adverse events.
Arm/Group | Clazakizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 2/8 | 2/8
Serious Adverse Events (participants affected / at risk) | 2/8 | 3/8
Other Adverse Events (participants affected / at risk) | 2/8 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clazakizumab (N=8) | Placebo (N=8)
Candida parapsilosis Fungemia (Infections and infestations) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 2 (2)
Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Multidrug-Resistant (MDR) Pseudomonas (Infections and infestations) | 1 (1) | 0 (0)
Pulseless Electrical Activity (PEA) Event (Cardiac disorders) | 0 (0) | 1 (1)
T12 Compression Fracture Secondary to Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Worsening Hypoxia (General disorders) | 1 (1) | 0 (0)
Worsening Kidney Function (Renal and urinary disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clazakizumab (N=8) | Placebo (N=8)
Acute Kidney Injury (AKI) (Renal and urinary disorders) | 0 (0) | 1 (1)
Delirium, multifactorial (Nervous system disorders) | 0 (0) | 1 (1)
Enterococcus faecalis Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Intermittent Atrial Fibrillation (AFib) with Labile Blood Pressure (Cardiac disorders) | 0 (0) | 1 (1)
Methicillin-susceptible staphylococcus aureus (MSSA) Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Paritonsillar Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Pseudomonas (Infections and infestations) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the small sample size, unable to assess statistical significance between the treatment and placebo group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT04348500/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT04348500/ICF_001.pdf